CLINICAL TRIAL: NCT07173491
Title: Effectiveness of Music-Based Interventions in Reducing Dental Anxiety During Restorative Dental Treatment
Brief Title: Music Therapy in Restorative Dentistry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Neslihan Celik, Assoc. Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TSA-2023-12101
Record Dates: First submitted 2025-09-02; First posted 2025-09-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Dental Anxiety
Keywords: restorative treatment; dental anxiety; music therapy

STUDY DESIGN:
Intervention Model Description: three groups with a control group
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- classical music group (Experimental): a music type used in the management of dental anxiety
  Interventions: Other: classical music group
- turkish music group (Experimental): a music type used in the management of dental anxiety
  Interventions: Other: turkish music group
- control (Placebo Comparator): no music therapy
  Interventions: Other: control

INTERVENTIONS:
Other: classical music group — classical music therapy with standard restorative treatment
  Arms: classical music group
Other: turkish music group — Turkish music therapy with standard restorative treatment
  Arms: turkish music group
Other: control — no music therapy with standard restorative treatment
  Arms: control

SUMMARY:
After administering a questionnaire to collect demographic data (including gender, age, education level, and frequency of dental visits) and MDAS scores, patients with an MDAS score of 10 or higher, indicating moderate to high dental anxiety, will be randomly allocated into three groups (n = 25 per group). Standard restorative treatment will be performed on the selected patients under music therapy.

DETAILED DESCRIPTION:
A single carpule of local anesthetic without vasoconstrictor will be administered to each patient using a disposable dental syringe. Following anesthesia, caries removal and cavity preparation will be performed. The restorative procedure will then commence. All procedures will be performed by the same clinician following a standardized protocol. Selective enamel etching will be performed with phosphoric acid for 30 seconds, followed by rinsing and gentle drying. Universal dental adhesive will be applied and polymerized according to the manufacturer's instructions. Subsequently, the prepared cavities will be restored with a resin composite, which will be light-cured for 20 seconds using an LED curing unit. Upon completion of finishing and polishing, the total duration of the restorative procedure will be recorded. Only one restoration will be performed for each patient.

Assessment of Physiological and Salivary Biomarkers In this study, systolic and diastolic blood pressure (SBP and DBP), oxygen saturation (SpO₂), heart rate (HR), salivary cortisol levels, salivary alpha-amylase (sAA) levels, and MDAS scores will be measured twice-once initially and once after the restorative procedure. Blood pressure will be recorded using a manual sphygmomanometer on the patients' right arms at heart level, and results will be expressed in mmHg. HR and SpO₂ will be measured with a finger-type portable pulse oximeter placed on the right index finger.

Unstimulated saliva samples will be collected from each participant just before and immediately after the procedure. Patients will be instructed to expectorate into sterile disposable tubes, ensuring the samples are free of blood contamination. To control for circadian fluctuations in cortisol and sAA levels, all samples will be collected between 9:00 and 12:00 a.m. The collected samples will be immediately stored at -80 °C until analysis.

A blinded researcher will perform all biochemical analyses after the completion of patient treatments. Samples will be thawed and centrifuged at 3,000 × g for 10 minutes. Cortisol concentrations will be determined using an enzyme-linked immunosorbent assay (ELISA) kit, while salivary alpha-amylase activity will be quantified with a colorimetric enzymatic assay. Absorbance values will be measured at a wavelength of 450 nm, and the results will be expressed in nanograms per milliliter (ng/ml) for cortisol and units for alpha-amylase.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy adults aged 18-40 years.
* Presence of D2 dentin caries confirmed by clinical and radiographic examination, characterized by radiolucency limited to the outer half of the dentin without pulpal or periapical pathology,
* Indication for single-session restorative treatment,
* Individuals with moderate-to-high dental anxiety according to the Modified Dental Anxiety Scale (MDAS), defined as a total score ≥10 (moderate: 10-18; high: ≥19).
* Ability and willingness to complete questionnaires and comply with study procedures.

Exclusion Criteria:

* deep dentin or pulpal involvement lesions, secondary caries, cracks, or fractured teeth,
* Acute or spontaneous dental pain, percussion sensitivity, or periapical pathology,
* Individuals with an MDAS total score ≤ 9 (no/low dental anxiety) were excluded.
* Hearing impairment or contraindications for music therapy,
* Psychiatric medication use or a diagnosed psychiatric disorder affecting anxiety response,
* Pregnant or breastfeeding individuals.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure (SBP) | at baseline and immediately after the restorative treatment
  Systolic blood pressure will be measured in a seated position using an automated sphygmomanometer. (Unit of Measure: mmHg)
Diastolic Blood Pressure (DBP) | at baseline and immediately after the restorative treatment
  Diastolic blood pressure will be measured in a seated position using an automated sphygmomanometer. (Unit of Measure: mmHg)
Oxygen Saturation (SpO₂) | at baseline and immediately after the restorative treatment
  Peripheral oxygen saturation will be assessed non-invasively using a finger pulse oximeter.
Heart Rate (HR) | at baseline and immediately after the restorative treatment
  Heart rate will be measured concurrently with blood pressure using an automated sphygmomanometer. (Unit of Measure: beats per minute (bpm))
Salivary Cortisol Levels | at baseline and immediately after the restorative treatment
  Salivary cortisol concentrations will be analyzed using an ELISA kit according to the manufacturer's protocol. (Unit of Measure: ng/mL)
Salivary Alpha-Amylase (sAA) Levels | At baseline and immediately after the restorative treatment
  Salivary alpha-amylase concentrations will be analyzed using an ELISA kit according to the manufacturer's protocol. (Unit of Measure: ng/mL)
Modified Dental Anxiety Scale (MDAS) Score | at baseline and immediately after the restorative treatment
  Anxiety levels will be assessed using the validated Modified Dental Anxiety Scale questionnaire. A 5-item anxiety scale; each item is rated 1-5 (Likert). The total score ranges from 5 to 25. Higher scores indicate greater dental anxiety (worse outcome). The outcome will be reported as change from baseline (Δ).

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk university, Faculty of dentistry, Department of restorative Dentistry clinics, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No